Steps for Epilepsy (StEpi)

NCT05359003

IRB Approved Date: 08MAY2024

# A FEASIBILITY STUDY OF A STEP-GOAL BASED PHYSICAL ACTIVITY INTERVENTION IN PEOPLE WITH EPILEPSY

Informed Consent Form to Participate in Research Halley Alexander, MD Principal Investigator

## **SUMMARY**

You are invited to participate in a research study. The purpose of this research is to help determine the best way to increase physical activity in people with epilepsy. You are invited to be in this study because you have epilepsy. Your participation in this research will involve 4 visits: (3 in-person visits and 1 telephone visit), plus telehealth visits as described below for your group, and last about 28 weeks.

Participation in this study will involve being randomized to either a control group or the intervention group. Both groups will wear a Garmin activity tracker and keep a study diary which will include recording information on seizures, sleep, and activity. The intervention group will participate in a 12-week walking physical activity intervention that is individualized to each participant's fitness level and abilities. This group will meet weekly with a coach who will monitor progress and provide exercise goals. At the end of the intervention period, the control group will be offered the opportunity to participate in the exercise program as well. All research studies involve some risks. A risk to this study that you should be aware of is the risk of falls or injuries related to starting an exercise program. There is a possibility that you may benefit from participation in this study.

Your participation in this study is voluntary. You do not have to participate in this study if you do not want to. There may be other choices available to you. Some other choices may include do nothing and continue your current care. You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study please contact the Principal Investigator at or

| If you have any questions, suggestions or concerns | s about your rights as a volunteer in this |
|---|---|
| research, contact the Institutional Review Board at | or the Wake Forest University |
| Health Sciences Research Subject Advocate at | • |

#### Introduction

You are invited to be in a research study. Research studies help scientists learn new information


Adult Consent Form

that may help other people in the future. You are being asked to be in this study because you have epilepsy. Your participation is voluntary. You do not have to be a part of this study if you do not want to. Please take your time in making your decision if you would like to join. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

## WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine whether a 12-week walking physical activity intervention, delivered by telehealth, is feasible in people with epilepsy. We will gather information on how you perform the physical activity, if you like or dislike the exercise program, and any issues you have completing the exercise. We will also look at whether this form of physical activity has effects on seizures, mood, stress, quality of life, and sleep.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

Up to 40 people at Wake Forest Baptist Health System will take part in this study. In order to identify the 40 subjects needed, we may need to screen as many as 3000 because some people will not qualify to be included in the study.

## WHAT IS INVOLVED IN THE STUDY?

All in-person study visits will occur either the Worrell Building, located on the Wake Forest University campus, or the Clinical Research Unit at Wake Forest Baptist Medical Center.

At your first visit, study staff will review the inclusion and exclusion criteria to ensure that you still qualify for the study. After reviewing the informed consent document (this document), you will have your vital signs taken. You will perform a 10 meter walk, which the staff will use to calculate your gait speed, in order to ensure that you are physically able to participate in the study. You will then be asked to provide basic information related to your medical history and your epilepsy.. You will be asked to perform some baseline assessments including a 6 minute walk, and a 10 minute resting heart rate measurement using a heart rate monitor. You will be asked to complete some questionnaires that will assess or ask questions about your mood, stress level, quality of life, medication side effects, goal setting, and exercise expectations. You will be given a Garmin Forerunner which will be setup with an application on your smartphone. You will be given a study diary, in which you will be asked to record your seizures, sleep, exercise, and any injuries, falls, or other issues that occur during the study period. This diary can be completed on paper but should be submitted daily electronically. You will then continue your normal habits for 4 weeks. It is important not to change your normal habits during this time. It is also important that you enter your diary results every day and wear your Garmin every day. If you do not do this, you will not be allowed to continue in the study.

At visit 2, you will undergo guided exercise testing on a treadmill. Then,

you will be <u>randomized</u> into one of the study groups described below. Randomization means that you are put into a group by chance. It is like flipping a coin, except in this case you have a 2:1


Adult Consent Form

odds of being in the exercise group. There are two groups you may be randomly assigned to in this study, one is the physical activity intervention group and the other is the education group.

If you are randomized into the study intervention group, this means you will participate in a 12-week physical activity program with a health coach. The physical activity will take place in your own home, using a daily step goal that will be assigned to you by your coach. You will meet with your coach weekly in a group format with other participants, which will be done remotely by video. You will also have weekly individual contact with your coach to review your *personal* progress and set new goals for the next week. This may be done by phone, video, or email, depending on your preference. In order to participate, you will need to have access to a smartphone and internet access or a cellular data plan for attending the virtual sessions. At the end of the 12-week intervention period, you will be encouraged to continue the physical activity/daily step goal on your own. We will evaluate your progress again at the end of another 12 weeks. During the second 12-week period, you will still fill out your diary and use your watch to track your physical activity, but you will NOT meet with a coach.

On the other hand, you may be assigned to the control group. Participating in the control groups means that you will continue your usual habits for 12 weeks. You will continue to wear the Garmin activity tracker but will not be given an exercise program. You will continue to log your daily seizure, sleep, and injuries/falls information in the study diary. You will be contacted by a study coordinator every 2 weeks for healthy living education. At the end of the 12 weeks, you will be offered free access to the exercise program if you want to participate.

Regardless of which group you are in, we ask you not to make changes to your seizure medications or seizure devices during this time. If changes are necessary as determined by your provider, then you may continue in the study, but please let us know. At the end of the 12-week intervention period, there will be an in-person follow up visit (Visit 3). At this visit, you will return to complete assessments and questionnaires similar to those that were given to you at the first visit. These include an exercise test, questionnaires, a 6-minute walk test, and another 10 minute heart rate measurement using a heart rate monitor. It may also include an exercise test like in Visit 1.

You will continue to complete your diary and wear your Garmin for another 12 weeks.

At the end of the study (about 28 weeks total), you will have a telephone visit (Visit 4) and will again answer a series of questionnaires and exit questions about being in the study will conclude at this time.

If you take part in this study, you will have the following tests and procedures. All of the following procedures will be done for research purposes only:

- Vital signs: Your blood pressure, heart rate, and weight will be taken at visits 1 and 3.
- 10 meter walk screen: At Visit 1, you will be asked to walk 10 meters. The staff will use to calculate your gait speed, in order to ensure that you are physically able to participate in the study. If you do not meet a certain speed, you will not be eligible to continue in the study.

Page **3** of **12**Adult Consent Form

- Collection of medical information: At Visit 1, your general information and medical information will be collected. This will include demographic information, and information about your epilepsy.
- Review seizure treatments: At all visits (Visits 1-4) your anti-seizure treatments will be reviewed, to ensure that there have been no changes during the study.
- Garmin Activity Tracker: You will receive a Garmin watch/activity tracker to wear on your wrist. It will be set up with de-identified information and a research account. You will be asked to wear this continuously while awake and asleep, only removing it while showering and while charging. Because we want to collect information about your sleep and activity, we recommend charging the device during periods of relative inactivity, such as when you are watching television or eating dinner, etc. Your personal information will not be recorded.
- ActivePAL4: This is an activity tracker that is worn on the thigh. Both groups will wear this for a 7-day period at the end of the baseline, intervention, and maintenance periods of the study.
- Study Diary: You will be asked to keep a study diary throughout the duration of the study period (28 weeks). You will record in this diary on a daily basis information regarding your seizures, sleep time, exercise, any fall/injuries, and hours wearing the Garmin device each day. You will submit this electronically and will get an email link every day to complete it.
- Questionnaires: At Visits 1, 3, and 4, you will be asked to complete a series of brief questionnaires regarding your mood, stress level, sleep quality, quality of life, and goal setting expectations. Some of these will be given in person and others will be done over the phone or sent to your email address to complete electronically.
- Heart-rate variability measurement: At Visits 1, 2 (optional if time permitting) and 3, we will measure an aspect of your heart rate called heart-rate variability. This simply requires you to sit quietly for 10 minutes while we record information with a heart monitor. It is not painful or invasive.
- 6 minute walk test: At Visits 1 and 3, you will be asked to complete a 6 minute walk test. The study staff will measure the distance that you are able to cover in 6 minutes. This is a measure of your physical fitness. You are allowed to rest during the test if you need to.
- Exercise Testing: You will undergo formal fitness testing on a treadmill in the presence of a physician. This will help determine your baseline level of fitness and your ability to safely participate in an exercise program.
- Exit Questions: At your last visit, we will ask you to answer a few short questions about your experience being in the study and any positive or negative feedback you have to help improve future studies.

#### If you are in the INTERVENTION group, you will also have:

- Weekly group coaching: This will be performed using video visits over the internet. You will be educated on how to access these. The entire visit will take roughly 1 hour.
- Weekly 1:1 session with coach: Performed by video, phone, or email, the coach will review
  with you the previous week's progress, troubleshoot any barriers, and give you new goals for
  the following week.
- Physical activity regimen: Your coach will give you a prescribed goal of daily steps for you each week. You can monitor these using your Garmin device.

 Adult Consent Form

- A post-intervention survey with questions asking how you liked, or didn't like, the physical activity program.
- Follow-up assessments at Visit 4 (week 28) performed remotely including many of the same questionnaires that you completed at Visits 1 and 3.

If you are in the control group, you will also have:

• Telephone health education every 2 weeks. This phone call will last  $\sim 20$  minutes.

As part of this research study, your group coaching sessions will be recorded. This is being done only so that the study staff can verify that the coaching sessions are being delivered correctly by the coach. These photographs/videotapes/audiotapes/recordings will be considered Protected Health Information if they contain information that identifies you. All Garmin tool data is deidentified and will only be viewed by members of the study team and will not be shared. You understand that you may request the photographing, filming, taping or recording be stopped at any time during the course of the research study, but doing so may affect your eligibility to remain in the research study. You should also understand that you will not be able to inspect, review, or approve the recordings.

These recordings will be destroyed once their use in this study is finished.

We can send copies of your test results to your personal physician if we find something concerning regarding your health and safety. Even if you do not wish to have any of your medical information sent to your physician, you can still participate in this research study.

Do you request that we send important medical findings from your study tests/exams to your personal physician?

| Γ | ] Yes | [ ] No | Initials |
|---|--------|--------|----------|
| L | J I es | [ ] NO | |

## HOW LONG WILL I BE IN THE STUDY?

You will be in the study for about 28 weeks.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first. There are no adverse risks to your health if you stop the study early.

## WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. Risks and side effects related to participation include:

Risks and side effects related to wearing the Garmin:

• There is minimal risk to wearing the Garmin device, which in rare cases may cause skin

Page **5** of **12** Adult Consent Form discomfort or irritation.

Risks and side effects related to the fitness test and exercise program: Likely

- Temporary shortness of breath and/or sweating from physical activity which is a normal physiological response but may be uncomfortable.
- Temporary muscle soreness or minor aches and pains after exercising.

#### Rare and Unexpected

- Severe shortness of breath or chest pain during the test, which may prompt further urgent or non-urgent work-up.
- Musculoskeletal injury causing more than temporary discomfort that requires further medical attention (such as ligament or tendon injury, muscle tear, muscle strain, etc.) Some injuries such as fractures or severe strains or tears could cause long-term physical discomfort.
- Worsening of seizures. For some people, exercise may trigger seizures. If you are in the intervention group and your seizure frequency worsens, we will not continue the intervention.

## Risks from Completing Questionnaires:

• Some of the questions asked may be upsetting, or you may feel uncomfortable answering them. If you do not wish to answer a question, you may skip it and go to the next question

Pregnant women are excluded from participation in this study. In the event you become pregnant while participating, you will be removed completely from the study immediately.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. In the group coaching, the importance of privacy and confidentiality of all information shared in the group session will be emphasized.

During the study, we ask that your anti-seizure medications and devices <u>are not changed during</u> the first 16 weeks of the study because we are trying to see if exercise can improve your epilepsy. You are probably used to your doctor making medication adjustments roughly every 3 months, so by participating in this study you may be prolonging this period of time by roughly 1 month. However, if medication changes are medically necessary, you can still continue in the study – please just let us know of any medication changes.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

As part of this study, you will be asked questions about your mood and passive suicidal thoughts. If we learn that you or someone else is in danger of harm, the study team is required to report that information to the proper authorities.

 Adult Consent Form There also may be other risks that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks to your health.

A Data Safety and Monitoring Committee, an independent group of experts, will be reviewing the data from this research throughout the study to identify possible safety issues to participants and to provide advice and recommendations on possible changes to the research study for the protection of participants.

## ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope the information learned from this study will benefit other people in the future. The benefits of participating in this study may be: improved sleep, lower stress, improved seizure control, improved mood, improved quality of life, and improved physical health.

Based on experience with exercise in animals with epilepsy and in people with other chronic diseases, researchers believe it may be of benefit to subjects with epilepsy. Because individuals respond differently to therapy, no one can know in advance if it will be helpful in your particular case.

## WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options:

- -continue current medical care as you normally would.
- -you may be eligible to participant in other research studies for epilepsy

The common standard of care is to continue increasing or adding anti-seizure medications, which have risks of side effects which vary according to the medication selected.

If your doctor wants you to consider epilepsy surgery, that work-up can still be pursued while you are in the study.

#### WHAT ARE THE COSTS?

All study costs, including any study products or procedures related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

## WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required or permitted by law, or necessary to protect the safety of yourself or others.

Your information may be provided to Federal and other regulatory agencies as required.


Adult Consent Form

By providing my email address, I give permission for Atrium Health, Wake Forest University Health Sciences, and their respective affiliated entities and representatives (including third-party agents if applicable) to send me information, reminders, and messages about the research study by email. I understand that these email messages may not be encrypted, and I understand and accept the risks that individuals not involved in the research study may be able to access unencrypted email messages. I also understand that email is not to be used for emergency situations.

## WILL YOU BE PAID FOR PARTICIPATING?

You will be paid \$200 if you complete all the scheduled study visits, but not intervention visits. If you withdraw for any reason from the study before completion you will be paid \$50 for each complete study visit.

To receive payment, you must provide your social security number, name and address so that we can comply with IRS (Internal Revenue Service) reporting requirements. When payments are reported to the IRS we do not let them know what the payment is for, only that you have been paid. If you do not wish to provide this information you can still take part in this study but you will not be paid.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

You will also be allowed to keep the Garmin device at the end of the study. If you do not complete the study, you will be asked to return the device.

## WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the Department of Neurology. The sponsor is providing money or other support to the researchers to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Wake Forest University Baptist Medical Center maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of injuries or illnesses to some participants in certain research studies. To the extent research insurance coverage is available under this policy, the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. To the extent research coverage is not available, you or your insurance company may be charged for the costs of medical care. You may receive care at Wake Forest University Baptist Medical Center and/or Atrium Health.

Page **8** of **12** Adult Consent Form If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Halley Alexander at or after hours call at the consent form.

## WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you] and/or [information we get from your medical records or other facilities about your health or behaviors is considered <a href="Protected Health Information">Protected Health Information</a>. The information we will collect for this research study includes: medical history including medical diagnoses, medications, imaging and other test results, employment information, age, gender, height, weight, zip code, phone number, email address, physical activity, fitness assessments and results from questionnaires regarding mood, sleep, quality of life, and exercise beliefs and goal setting.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study may be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with the health care operations of Atrium Health, Wake Forest University Health Sciences, and their respective affiliated entities.

We will take steps to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and Atrium Health Facilities; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy

 Adult Consent Form regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs, videotapes, audiotapes or other recorded media which are identify you unless we you're your written authorization.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to your medical record for verification of clinical trial procedures or data to the extent permitted by other applicable laws. These monitors, auditors, and other individuals are also required to maintain the confidentiality of your protected health information.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for at least six years after the study is finished. At that time any research information not already in your medical record will either be destroyed or it will be deidentified.

Any research information entered into your medical record will be kept for as long as your medical record is kept by the Medical Center. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Halley Alexander, MD that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form, you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Atrium Health, Wake Forest University Health Sciences, or their respective affiliated entities will indicate that you are

 Adult Consent Form enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. Authorization to access this part of the medical record will only be available to people who have a need to know this information in order to perform their job-related duties. If you are not a patient of these health care facilities, a medical record will be created for you anyway to provide access to this important information to providers in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other clinically relevant medical reports created as a result of your participation in the research study may be entered into the computer systems of Atrium Health, Wake Forest University Health Sciences, and/or their respective affiliated entities. These results and reports will be kept secure in compliance with applicable laws, with permission to access this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A medical record will be created for all study participants seen on-site and if a medical record doesn't already exist. Information about your participation in the study will be placed in the medical record, along with any routine medical test results that were obtained as part of this study.

## WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped. Information that identifies you may be removed from the data or specimens that are collected as part of this study and could be used for future research or shared with others without additional consent.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Halley Alexander, MD at or after hours at ...

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like

 Adult Consent Form

| to discuss problems or concerns, have questions or additional information, you should contact the Charlesearch Subject Advocate at | - | | |
|---|---|---|---|
| You will be given a copy of this signed consent for | rm. | | |
| SIGNATURES | | | |
| If you agree to receiving text messages, please pro agree, you understand and accept the risks associate may apply. You will receive text messages about statement DESCRIPTION OF CONTENT]. If you prefer not these communications by email (with your agreem number with another person, there is a chance they | ted with text message<br>tudy related visits a<br>t to receive text mest<br>tent), mail, or phone | ging and that da<br>nd procedure [lassages, you will<br>be. If you share y | ta charges INSERT receive |
| YES, preferred phone number | | | |
| NO | | | |
| Participant Signature: | Date: | Time: | am pm |
| I agree to take part in this study. I authorize the use described in this consent and authorization form. Privacy Notice, I may request one or one will be mask questions about being in this study and have the consent and authorization form, I am not releasing sponsor, the institution or its agents from liability in | If I have not already<br>nade available to me<br>lose questions answ<br>or agreeing to relea | received a cope. I have had a ered. By signi | y of the chance to ng this |
| Subject Name (Printed): | | | |
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent (Printed): | | | |
| Person Obtaining Consent: | Date: | Time: | am pm |

 Adult Consent Form